CLINICAL TRIAL: NCT02131935
Title: Impaired Peripheral Endothelial Function as Assessed by Digital Reactive Hyperemia Peripheral Arterial Tonometry and Risk of In-Stent Restenosis
Brief Title: Impaired Peripheral Endothelial Function and In-stent Restenosis
Status: Completed | Type: Observational
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Kenichi Tsujita, MD, PhD, Assistant Professor, Kumamoto University
Other Study IDs: 1120
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ISR Group: Patients Group Experienced In-Stent Restenosis (ISR)
- Non-ISR: Patients Group Without in-stent restenosis (ISR)

SUMMARY:
The investigators assessed the hypothesis that whether RH-PAT index (RHI) as a marker of endothelial dysfunction could predict occurrence of ISR after percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
This is a prospective observational study of all consecutive patients with coronary artery disease (CAD) treated with PCI at Kumamoto University Hospital between January 2010 and September 2012. Inclusion criteria consisted of patients who were symptomatic for myocardial ischemia and who were undergoing stent implantation for significant CAD.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria consisted of patients who were symptomatic for myocardial ischemia and who were undergoing stent implantation for significant CAD.

Exclusion Criteria:

* Exclusion criteria were balloon angioplasty only without stent deployment, death during hospitalization, and patients who had comorbidities affected RH-PAT results such as hemodialysis, advanced cancer, after surgery of breast cancer, dementia, collagen disease, and not performing RH-PAT with uncertain reason.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patient sampling This is a prospective observational study of all consecutive patients with coronary artery disease (CAD) treated with PCI at Kumamoto University Hospital between January 2010 and September 2012. Inclusion criteria consisted of patients who were symptomatic for myocardial ischemia and who were undergoing stent implantation for significant CAD.
Sampling Method: Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Presence or absence of in-stent restenosis | within 1 year
  Based on the Japanese clinical routine, follow-up (F/U) angiography will be performed at six and nine months after PCI with bare-metal stent (BMS) and drug-eluting stent (DES), respectively. ISR was defined as percent diameter stenosis >50% at F/U angiography assessed by quantitative coronary angiography.

SECONDARY OUTCOMES:
Endothelial Function | within 1 year
  Fingertip reactive hyperemia peripheral arterial tonometry (RH-PAT) is a new device that provides noninvasive, automatic, and quantitative evaluation of endothelial dysfunction with low intra- and inter-observer variability. We assess the hypothesis that whether RH-PAT index (RHI) as a marker of endothelial dysfunction could predict occurrence of ISR after percutaneous coronary intervention (PCI). RHI will be measured using Endo-PAT2000 (Itamar Medical, Caesarea, Israel) before PCI (initial RHI) and at follow-up angiography (F/U RHI) in consecutive patients who had successful PCI in de novo coronary lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, MD, PhD, Study Chair — Kumamoto University
Locations (1):
- Kumamoto University, Kumamoto, Kumamoto, Japan

REFERENCES:
- [Derived] Komura N, Tsujita K, Yamanaga K, Sakamoto K, Kaikita K, Hokimoto S, Iwashita S, Miyazaki T, Akasaka T, Arima Y, Yamamoto E, Izumiya Y, Yamamuro M, Kojima S, Tayama S, Sugiyama S, Matsui K, Nakamura S, Hibi K, Kimura K, Umemura S, Ogawa H. Impaired Peripheral Endothelial Function Assessed by Digital Reactive Hyperemia Peripheral Arterial Tonometry and Risk of In-Stent Restenosis. J Am Heart Assoc. 2016 Jun 17;5(6):e003202. doi: 10.1161/JAHA.116.003202. PMID 27317348